CLINICAL TRIAL: NCT02359552
Title: A 24-week, Three-site, Randomized, Double Blind, Placebo Controlled, Parallel Group, Proof-of-concept Study to Evaluate Rasagiline in the Regional Brain Metabolism on FDG PET in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Rasagiline Rescue in Alzheimer's Disease Clinical Trial
Acronym: R2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-519
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be randomized in 1:1 ratio to receive Rasagiline or the matching placebo 24-week double blind treatment.
  Subjects will take one 0.5 mg Rasagiline tablet or the matching placebo once a day on Baseline (Day 1) through Week 4. The dose will be titrated up to one 1 mg tablet or the matching placebo once a day starting on Week 5 until the Week 28 (end of treatment visit).
  Interventions: Drug: Placebo
- Rasagiline (Active Comparator): Subjects will be randomized in 1:1 ratio to receive Rasagiline or the matching placebo 24-week double blind treatment.
  Subjects will take one 0.5 mg Rasagiline tablet or the matching placebo once a day on Baseline (Day 1) through Week 4. The dose will be titrated up to one 1 mg tablet or the matching placebo once a day starting on Week 5 until the Week 28 (end of treatment visit).
  Interventions: Drug: Rasagiline

INTERVENTIONS:
Drug: Rasagiline
  Arms: Rasagiline
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase II, randomized, double blind, placebo controlled, parallel group, proof of concept three-site study, to evaluate the effect of Rasagiline in the regional brain metabolism on 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG-PET).

DETAILED DESCRIPTION:
The study consists of two phases: a 24 week double blind placebo controlled treatment period and a 4 week follow up period. Patients will be randomized in a 1: 1 ratio at baseline to receive either Rasagiline or matching placebo

The study drug will be given as 0.5 mg dose once daily for the 4 weeks, then increases to 1 mg daily for the next 20 weeks. A total of 50 subjects will be enrolled: 25 will receive Rasagiline and 25 will receive matching placebo for the 24-week treatment period.

Primary objective is to determine if exposure to 1 mg of Rasagiline daily is associated with improved regional brain metabolism in the treatment group compared to the placebo group in Alzheimer's Disease patients

ELIGIBILITY:
Inclusion Criteria:

* Males or females 50 to 90 of age inclusive.
* Diagnosis of probable AD (NINCDS-ADRDA criteria)
* Positive fluoro-deoxyglucose PET ([18F]-FDG PET) scan compatible with AD as determined by the ADM Diagnostics LLC (ADMdx) Criteria at screening
* Mini Mental Status Exam = 12 - 22 (inclusive)
* Must have a study partner who is able and willing to comply with all required study procedures.
* Have at least eight years of education and should have previously (in pre-AD condition) been capable of reading, writing, and communicating effectively with others in English.
* If receiving therapy with a cholinesterase inhibitor and/or memantine, the dose of these agents has been stable for at least 3 months prior to screening

Exclusion Criteria:

* Any non-AD neurological disease
* MRI findings indication of a non-AD diagnosis
* Screening laboratory studies that are 1.5 times above or below the highest and lowest range of normal for each test respectively
* History of melanoma; history of malignancy within the past five years with the exception of basal cell or squamous cell cancer, in-situ cervical cancer, or localized prostate cancer

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2019-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Cummings, MD, ScD, Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (3):
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Cleveland Clinic Lakewood Hospital, Lakewood, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Galasko D, Bennett D, Sano M, Ernesto C, Thomas R, Grundman M, Ferris S. An inventory to assess activities of daily living for clinical trials in Alzheimer's disease. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S33-9. PMID 9236950
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited based on physician referral from three Cleveland Clinic sites between May 2015 and January 2018
Pre-assignment Details: Of 96 screened participants, 50 met inclusion criteria and were enrolled and randomized to treatment.
Groups:
- Placebo: Subjects will be randomized in 1:1 ratio to receive Rasagiline or the matching placebo 24-week double blind treatment.
  Subjects will take one 0.5 mg Rasagiline tablet or the matching placebo once a day on Baseline (Day 1) through Week 4. The dose will be titrated up to one 1 mg tablet or the matching placebo once a day starting on Week 5 until the Week 28 (end of treatment visit).
  Placebo
- Rasagiline: Subjects will be randomized in 1:1 ratio to receive Rasagiline or the matching placebo 24-week double blind treatment.
  Subjects will take one 0.5 mg Rasagiline tablet or the matching placebo once a day on Baseline (Day 1) through Week 4. The dose will be titrated up to one 1 mg tablet or the matching placebo once a day starting on Week 5 until the Week 28 (end of treatment visit).
  Rasagiline
Period: Overall Study
Arm/Group | Placebo | Rasagiline
Started | 25 | 25
Completed | 22 | 21
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rasagiline | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.44 (7.12) | 74.72 (7.35) | 74.08 (7.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 14 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Alzheimer's Disease Assessment Scale - Cognitive 11 score [Mean (Standard Deviation); unit: units on a scale] — The ADAS-Cog 11 is a psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis. A higher score indicates worse impairment. Scores range test from 0 (best) to 70 (worse). We used total ADAS-Cog 11 scores, which is a sum of individual subscales.
  units on a scale | 27.96 (10.53) | 23.2 (6) | 25.58 (8.81)
Mini Mental Status Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The MMSE is a brief, frequently used screening instrument for AD drug studies. The MMSE evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two overlapping pentagons. A lower score indicates more cognitive impairment. The highest score is 30.
  units on a scale | 19.04 (4.61) | 21.24 (3.54) | 20.14 (4.21)
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) score [Mean (Standard Deviation); unit: units on a scale] — The ADCS-ADL is an activities-of-daily-living inventory developed by the ADCS to assess functional performance in participants with AD. Using a structured interview format, study partners are queried as to whether participants attempted each item in the inventory during the past 4 weeks and their level of performance. The ADCS-ADL provides a total score from 0-78, with a lower score indicating greater severity.
  units on a scale | 58.2 (11.1) | 61.88 (8.44) | 60 (9.96)
Neuropsychiatric Inventory (NPI) score [Mean (Standard Deviation); unit: units on a scale] — The behavioral outcome measure for this trial is the Neuropsychiatric Inventory (NPI). The NPI evaluates both the frequency and severity of 10 neuropsychiatric disturbances. Frequency assessments range from 1 (occasionally, less than once per week) to 4 (very frequently, once or more per day or continuously) as well as severity (1=mild, 2=moderate, 3=severe). The overall score is calculated by summing the severity and frequency of the subscale measures. The range of scores is from 0-40. A score of 0 indicates no neuropsychiatric disturbance while a score of 40 indicates severe disturbance.
  units on a scale | 8.28 (8.97) | 7.62 (7.61) | 7.96 (8.25)
digit span [Mean (Standard Deviation); unit: units on a scale] — The Digit Span consists of repetition of increasing long strings of digits presented at 1 per second as read by the examiner and repeated by the subject.The score is the maximum number of digits the patient can repeat until they fail twice in a row. The reverse digit span is identical to the forward digit span except that the patient repeats the presented digits in reverse order. The score is the maximum number of digits the patient can repeat in reverse order until they fail twice in a row. Each correct response is worth one point with a maximum total score of 28. A higher score is better.
  units on a scale | 11.76 (3.23) | 13.08 (2.75) | 12.42 (3.04)
Controlled Oral Word Association Test (cowat) score [Mean (Standard Deviation); unit: units on a scale] — Study participants are instructed, "I want to see how many words you can say beginning with a certain letter in one minute." The study participant's responses are recorded on the worksheet. Study participants are then given an additional one minute for each of two different letters using similar instructions. The score is the total number of acceptable words for the three trials combined. A higher score represents better performance. The range of scores is from 0-100.
  units on a scale | 21.16 (13.16) | 26.72 (12.6) | 23.94 (13.06)
Quality of Life - Alzheimer's Disease (QoL-AD) [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life in Alzheimer's Disease (QoL-AD) is a commonly used 13 item quality of life (QoL) scale that assesses items specific to QoL in patients with cognitive impairment. It is administered to the research partner who answers for the patient. Points are assigned to each item as follows: poor = 1, fair = 2, good = 3, excellent = 4.The total score is the sum of all 13 items. The range of score is 0 to 52. A score of 0 indicates severe impairment and a score of 52 indicating no impairment.
  units on a scale | 39.58 (5.24) | 36.73 (5.35) | 38.22 (5.43)

OUTCOME MEASURES:

1. Primary Outcome: Change in Regional Glucose Metabolism Between Week 24 and Baseline as Measured by 18F-2-fluoro-2-deoxy-D-glucose Positron Emission Tomography (FDG-PET).
Description: The primary outcome measure is the change from baseline to week 24 in FDG-PET as measured by Standard Uptake Units Regional (SUVR) in several pre-specified brain regions including the medial temporal, lateral temporal, posterior cingulate - precuneus, inferior parietal, middle frontal, anterior cingulate, and striatum. The SUVR change was calculated by subtracting the value at 24 weeks from baseline values. Negative values indicate increased hypometabolism (i.e. worsening of cell function).
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 25 | 25
SUVR
  Middle Frontal | -0.032 (0.030) | -0.011 (0.030)
  Anterior Cingulate | -0.020 (0.021) | -0.003 (0.026)
  Superior Frontal | -0.016 (0.022) | -0.003 (0.018)
  Striatum | -0.024 (0.029) | -0.002 (0.028)
  Medial Temporal | -0.015 (0.034) | -0.010 (0.034)
  Lateral Temporal | -0.020 (0.029) | -0.016 (0.024)
  Post Cingulate - Precuneus | -0.017 (0.023) | -0.016 (0.018)
  Inferior Parietal | -0.025 (0.029) | -0.018 (0.022)

2. Secondary Outcome: Change in ADAS-Cog 11 (Alzheimer's Disease Assessment Scale - Cognitive 11) Score
Description: The ADAS-Cog 11 (Alzheimer's Disease Assessment Scale - Cognitive 11) is a psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis. A higher score indicates more impairment. Scores from the original portion of the test range from 0 (best) to 70 (worse). We used total ADAS-Cog 11 scores, which is a sum of individual subscales. We calculated the change by subtracting the ADAS Cog score at week 24 from baseline score. A positive change indicates cognitive worsening.
Time Frame: Mean change in scores from baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 25 | 25
score on a scale | 2.76 (4.3) | 1.81 (4.43)

3. Secondary Outcome: Change in MMSE (Mini Mental Status Examination) Score
Description: Measure Description: The MMSE (Mini Mental Status Examination) is a brief, frequently used screening instrument for AD drug studies. The MMSE evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two overlapping pentagons. A lower score indicates more cognitive impairment. The highest score is 30, range is between 0 (severe impairment) and 30 (cognitively normal). We calculated the change in scores by subtracting week 24 score from baseline. A negative score indicates clinical worsening.
Time Frame: Mean change in scores from baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 25 | 25
score on a scale | -1.14 (2.27) | -0.65 (2.48)

4. Secondary Outcome: Change in ADCS-ADL (Alzheimer's Disease Cooperative Study-Activities of Daily Living) Score
Description: Measure Description: The ADCS-ADL (Alzheimer's Disease Cooperative Study-Activities of Daily Living) is an activities-of-daily-living inventory developed by the ADCS to assess functional performance in participants with AD. Using a structured interview format, study partners are queried as to whether participants attempted each item in the inventory during the past 4 weeks and their level of performance. The ADCS-ADL provides a total score from 0-78, with a lower score indicating greater severity. We calculated change by subtracting scores on week 24 test from the baseline score. A negative score indicates worsening ability to complete ADLs.
Time Frame: Mean change in scores from baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 25 | 25
score on a scale | -3.23 (6.71) | -3.75 (7.27)

5. Secondary Outcome: Change in NPI (Neuropsychiatric Inventory) Score
Description: Measure Description: The behavioral outcome measure for this trial is the NPI (Neuropsychiatric Inventory). The NPI evaluates both the frequency and severity of 10 neuropsychiatric disturbances. Frequency assessments range from 1 (occasionally, less than once per week) to 4 (very frequently, once or more per day or continuously) as well as severity (1=mild, 2=moderate, 3=severe). The overall score is calculated by summing the severity and frequency of the subscale measures. The range of scores is 0-40. A score of 0 indicates no behavioral impairment and a score of 40 indicates severe behavioral impairment. We calculated change by subtracting Week 24 scores from baseline scores. A positive change indicates behavioral worsening.
Time Frame: Mean change in scores from baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 25 | 25
score on a scale | 2 (7.18) | 0.2 (6.79)

6. Secondary Outcome: Change in Digit Span
Description: Measure Description: The Digit Span consists of repetition of increasing long strings of digits presented at 1 per second as read by the examiner and repeated by the subject.The score is the maximum number of digits the patient can repeat until they fail twice in a row. The reverse digit span is identical to the forward digit span except that the patient repeats the presented digits in reverse order. The score is the maximum number of digits the patient can repeat in reverse order until they fail twice in a row. Each correct response is worth one point with a maximum total score of 28. A higher score is better. We calculated change by subtracting week 24 score from baseline score. A negative score indicates worse performance over the course of study.
Time Frame: Mean change in scores from baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 25 | 25
score on a scale | -1.18 (1.92) | -0.29 (3.08)

7. Secondary Outcome: Change in COWAT (Controlled Oral Word Association Test) Score
Description: Measure Description: Study participants are instructed, "I want to see how many words you can say beginning with a certain letter in one minute." The study participant's responses are recorded on the worksheet. Study participants are then given an additional one minute for each of two different letters using similar instructions. The score is the total number of acceptable words for the three trials combined. A higher score represents better performance.
  Responses are then judged for their acceptability (example for the use of proper nouns, numbers, repetitions and stem word with a different ending). The score is the total number of acceptable words for the three trials combined. A higher score represents better performance. We calculated change by subtracting week 24 scores from baseline scores. A negative score indicates worse performance.
Time Frame: Mean change in scores from baseline to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 25 | 25
score on a scale | -1.09 (6.31) | 0.62 (5.55)

8. Secondary Outcome: Change in QoL-AD (Quality of Life - Alzheimer's Disease) Score
Description: Measure Description: The QoL-AD (Quality of Life - Alzheimer's Disease) is a commonly used 13 item QoL scale that assesses items specific to QoL in patients with cognitive impairment. It is administered to the research partner with answers for the patient. Points are assigned to each item as follows: poor = 1, fair = 2, good = 3, excellent = 4.The total score is the sum of all 13 items. The range of score is from 0-52. We calculated the change by subtracting the scores on week 24 score from baseline. A negative value indicates worsening quality of life.
Time Frame: This assessment will be performed at the Baseline and Week 24 visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 25 | 25
score on a scale | -1.95 (3.28) | 1.11 (3.77)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected following signing of consent to completion of study week 28 (from May 2016 to August 2018). At each point of contact the research coordinator and PI collected data regarding any new symptoms or laboratory changes.
Arm/Group | Placebo | Rasagiline
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 4/25 | 1/25
Other Adverse Events (participants affected / at risk) | 15/25 | 16/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Rasagiline (N=25)
confusion (Psychiatric disorders) | 1 (1) | 0 (0)
delusions (Psychiatric disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
stroke (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Rasagiline (N=25)
Abnormal UA (Renal and urinary disorders) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 2 (2)
Delusions (Psychiatric disorders) | 3 (3) | 3 (3)
Elevated blood pressure (Vascular disorders) | 2 (2) | 3 (3)
Elevated Thyroid Stimulating Hormone (Endocrine disorders) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Rash/skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT02359552/Prot_000.pdf
  • Statistical Analysis Plan (2014-09-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT02359552/SAP_001.pdf